CLINICAL TRIAL: NCT05268874
Title: The Effect of Clavipectoral Fascia Plane Block on Pain Management and Patient Satisfaction Following Clavicle Surgery: Randomized, Prospective Study
Brief Title: The Effectiveness of Clavipectoral Fascia Plane Block for Clavicle Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medipol University (Other)
Responsible Party: Principal Investigator, Bahadir Ciftci, Principal Investigator, Medipol University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Mugla Sitki Kocman University
Record Dates: First submitted 2022-02-10; First posted 2022-03-07 (Actual); Last update posted 2022-09-19 (Actual); Status verified 2022-09

CONDITIONS: Clavicle Fracture; Clavicle Injury
Keywords: Clavicle surgery; Postoperative pain management; Clavipectoral fascia plane block

STUDY DESIGN:
Intervention Model Description: 38 patients aged 18-65 years old with American Society of Anesthesiologists (ASA) classification I-II and scheduled for clavicle surgery will be included in the study. Patients will be randomly divided into two groups (Group Clavipectoral and Group Control) including 19 patients each, before entering the operating room.
Who Masked: Participant, Outcomes Assessor
Masking Description: Outcomes Assessor and participant will be blinded to the study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group Clavipectoral = Clavipectoral block group (Active Comparator): Patients will be administered ibuprofen 400 mgr IV every 8 hours in the postoperative period. Postoperative patient evaluation will be performed by a pain nurse blinded to the procedure. Tramodol will be performed for rescue analgesia.
  Interventions: Other: Clavipectoral block
- Group Control = Control group (No Intervention): Patients will be administered ibuprofen 400 mgr IV every 8 hours in the postoperative period. Postoperative patient evaluation will be performed by a pain nurse blinded to the procedure. Tramodol will be performed for rescue analgesia.

INTERVENTIONS:
Other: Clavipectoral block — Clavipectoral block will be performed with patients in the supine position. The probe will be placed on the anterior border of the medial third (or on the proximal or distal end, according to the localization of the fracture) of the clavicle. A 22-gauge, 50 mm block needle will be inserted in a caudal to cephalic direction, the periosteum of the clavicle and the surrounding fascia will be visualized, 30 ml of 0.25% bupivacaine will be injected between these two layers. The local anesthetic spread to medial and lateral third of the clavicle will be seen.
  Arms: Group Clavipectoral = Clavipectoral block group

SUMMARY:
Clavipectoral fascia plane block (CPB). CPB was defined by Valdes in 2017 firstly. It may be used for postoperative analgesia after clavicle surgery. In the literature, data about CPB is so limited, however it seems a good option for pain management after clavicle fracture.

The aim of this study is to evaluate the efficacy of the ultrasound-guided CPB for postoperative analgesia management and patient satisfaction in patients underwent clavicle surgery.

DETAILED DESCRIPTION:
Clavipectoral fascia plane block (CPB) was defined by Valdes in 2017 firstly. It may be used for postoperative analgesia after clavicle surgery. The clavipectoral fascia covers the clavicular site of the pectoralis major muscle. It provides the potential interfascial space between the clavicle and the pectoralis major muscle. CPB provide effective analgesia after clavicle surgery. It is also easy to perform. With this advantage and its analgesic effectiveness for clavicle surgery, CPB may be an alternative to interscalene brachial plexus block. However, randomized clinical efficacy trials are needed to investigate the effectiveness of CPB for clavicle fractures. In the literature, data about CPB is so limited, however it seems a good alternative to brachial plexus block for pain management after clavicle fracture

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anesthesiologists (ASA) classification I-II
* Scheduled for clavicle surgery under general anesthesia

Exclusion Criteria:

* bleeding diathesis,
* anticoagulation,
* thorax wall abnormalities
* study drug allergy,
* infection at the block area,
* pregnancy or lactation,
* patients who do not accept the procedure

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2022-03-18 (Actual); Primary Completion 2022-09-16 (Actual); Study Completion 2022-09-16 (Actual)

PRIMARY OUTCOMES:
Postoperative pain scores (NRS) | Postoperative 24 hours period
  The primary outcome is the NRS at postoperative 8th hour

SECONDARY OUTCOMES:
The use of rescue analgesia (number of participants and rate of tramodol using) | Postoperative 24 hours period
  Tramodol using
Patient satisfaction | Postoperative at 24th hour
  Patient satisfaction will be evaluated with seven item Likert scala

CONTACTS AND LOCATIONS:
Locations (1):
- Mugla Sıtkı Kocman University Hospital, Muğla, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
We will not plan to share IPD

REFERENCES:
- [Background] Atalay YO, Mursel E, Ciftci B, Iptec G. Clavipectoral Fascia Plane Block for Analgesia after Clavicle Surgery. Rev Esp Anestesiol Reanim (Engl Ed). 2019 Dec;66(10):562-563. doi: 10.1016/j.redar.2019.06.006. Epub 2019 Nov 11. No abstract available. English, Spanish. PMID 31727320
- [Background] Atalay YO, Ciftci B, Ekinci M, Yesiltas S. The effectiveness of clavipectoral fascia plane block for analgesia after clavicle surgery: a report of five cases. Minerva Anestesiol. 2020 Sep;86(9):992-993. doi: 10.23736/S0375-9393.20.14503-6. Epub 2020 May 18. No abstract available. PMID 32420714
- [Background] Kukreja P, Davis CJ, MacBeth L, Feinstein J, Kalagara H. Ultrasound-Guided Clavipectoral Fascial Plane Block for Surgery Involving the Clavicle: A Case Series. Cureus. 2020 Jul 8;12(7):e9072. doi: 10.7759/cureus.9072. PMID 32782888
- [Background] Magalhaes J, Segura-Grau E. Single puncture clavipectoral fascial block as a potential effective analgesic strategy for clavicle surgery. J Clin Anesth. 2020 Dec;67:110062. doi: 10.1016/j.jclinane.2020.110062. Epub 2020 Sep 23. No abstract available. PMID 32979611